CLINICAL TRIAL: NCT06667960
Title: A Phase 1/2, Multicenter, Open Label, Dose Escalation & Dose Expansion Study of JK06, a 5T4 Antibody Drug Conjugate, in Patients With Unresectable Locally Advanced or Metastatic Cancer
Brief Title: Study of JK06 in Patients With Unresectable Locally Advanced or Metastatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Salubris Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JK06.1.01
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose Escalation phase will use a 3+3 design with enrollment of 3 patients per cohort and expansion to 6 patients in the event of a DLT. The Dose Escalation phase will determine the MTD/recommended phase 2 dose (RP2D) for Cohort Expansion.
  In the Cohort Expansion phase of the study, up to 3 parallel cohorts of patients with specific tumor types, and a cohort of mixed solid tumors will simultaneously enroll and be treated to further characterize the safety, tolerability, PK, pharmacodynamics, and anti-tumor activity of JK06
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Escalating repeated doses of JK06 administered intravenously. A cycle of treatment is defined as 21 days.
  Interventions: Drug: JK06
- Dose Expansion (Experimental): The RP2D/OBD of JK06 determined by the Escalation arm. A cycle of treatment is defined as 21 days.
  Interventions: Drug: JK06

INTERVENTIONS:
Drug: JK06 — Biparatopic anti-5T4 antibody

SUMMARY:
This is a Phase 1/2, open-label, multi-center, first-in-human, dose escalation and cohort expansion study evaluating multiple doses and schedules of intravenously administered JK06 in patients with unresectable locally, advanced or metastatic cancer.

DETAILED DESCRIPTION:
This Phase 1/2, open label, dose escalation and cohort expansion study is designed to evaluate and characterize the safety, tolerability, PK, pharmacodynamics, immunogenicity, and preliminary anti-tumor activity of JK06 administered intravenously (IV) in patients with unresectable, locally advanced, or metastatic cancer. The study consists of a Dose Escalation phase to determine the MTD/recommended phase 2 dose (RP2D) of JK06, followed by a Cohort Expansion phase to further define the safety and initial efficacy of JK06 in tumor specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old. 2. Signed informed consent and willing and able to comply with study procedures and scheduled visits.

  3. For Dose Escalation, patients with histologically diagnosed unresectable, locally advanced, or metastatic solid tumors.

  4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1. 5. Life expectancy ≥ 12 weeks. 6. Measurable disease as per RECIST 1.1 criteria and documented by CT and/or MRI.

Note: lesions treated previously with radiation must demonstrate clear evidence of radiographic progression since the completion of prior radiotherapy and prior to study enrollment.

7. Acceptable laboratory parameters:

* Albumin ≥ 2.8 g/dL.
* Platelet count ≥ 100, 000.
* Hemoglobin ≥ 9.0 g/dL.
* Absolute neutrophil count ≥ 1,500/μL.
* ALT/AST ≤ 3.0 times ULN.

  - ALT/AST ≤ 5 × ULN for patients with liver metastases.
* Total bilirubin ≤ 1.5 ULN or ≤ 3 x ULN for patients with Gilbert's disease.
* Direct bilirubin ≤ 1.5 ULN for patients with total bilirubin > 1.5 ULN.
* Creatinine ≤ 1.8 mg/dL.

  * Or calculated/measured creatinine clearance > 30 mL/minute. 8. Identification of an archival tumor sample (i.e., tissue block (formalin-fixed paraffin-embedded [FFPE]) or a series of approximately 10-15 slides).

    9. Consent to pre-treatment fresh tumor biopsy for patients enrolled in the back-fill part of Dose Escalation and all eligible patients enrolled in Cohort Expansion.

    10. Women of childbearing potential (WOCBP) not surgically sterilized and between menarche and 1 year post menopause must have a negative serum or urine pregnancy test.

    11. Treated central nervous system (CNS) metastases 12. Must be willing and able to comply with clinic visits and procedures outlined in the study protocol.

    13. Concurrent use of hormones for breast cancer or for non-cancer related conditions (e.g., insulin for diabetes, hormone replacement therapy) is acceptable. Bisphosphonates or RANK-L inhibitors or analogues are permitted for supportive care of patients with bone metastases.

Exclusion Criteria:

1. Patients with symptomatic or unstable CNS primary tumor or metastases and/or carcinomatous meningitis. Patients with documented treated CNS metastases stable for at least 4 weeks may be enrolled at the discretion of the investigator.
2. Major surgery within 6 weeks from treatment initiation.
3. Clinically significant cardiovascular/vascular disease ≤ 6 months before first dose.
4. Clinically significant gastrointestinal disorders.
5. Clinically significant pulmonary compromise requiring supplemental oxygen use.
6. Grade 2 or greater peripheral neuropathy at time of study entry.
7. Vaccination with any live virus vaccine within 4 weeks prior to the initiation of study drug administration. Inactivated annual influenza vaccination is allowed.
8. Known hypersensitivity to JK06 or any excipient.
9. Second primary invasive malignancy not in remission for ≥ 1 year. Exceptions include non-melanoma skin cancer, cervical carcinoma in situ, resected melanoma in situ, or any malignancy considered to be indolent and never required therapy.
10. Any serious underlying medical or psychiatric condition that would preclude understanding and rendering of informed consent or impair the ability of the patient to receive or tolerate the planned treatment.
11. Recent or ongoing serious infection.
12. Prior systemic anti-cancer treatment:

    * For cytotoxic chemotherapy, small molecule inhibitors, radiation, or similar investigational treatments, ≤ 2 weeks or 5 half-lives, whichever is shorter.
    * For monoclonal antibodies or similar experimental therapies: ≤ 3 weeks or 5 half-lives, whichever is shorter.
    * Antibody drug conjugates and radioimmunoconjugates or other similar experimental therapies ≤ 6 weeks or 5 half-lives, whichever is shorter.
13. Ascites or pleural effusions requiring large volume para- or pleurocentesis within 4 weeks of treatment initiation.
14. Pregnant or nursing.
15. Therapeutic anticoagulation for a thromboembolic event that occurred within 3 months of dosing; prophylactic anticoagulation is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Dose-Finding | From First Patient Dosed to end of Escalation, up to 14 months.
  Determination of the maximum-tolerated dose/recommended Phase 2 dose.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | First treatment through 28 days after last dose of treatment or End of Treatment [EOT] visit, whichever is later.
  Incidence, nature, and severity of treatment-emergent adverse events [TEAEs]. Defined as any AE that occurs during the treatment period (i.e., after any treatment) and up to 28 days after the last dose of study treatment.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Screening date through 28 days after last dose of treatment or End of Treatment [EOT] visit, whichever is later.
  Incidence, nature, and severity of Serious Adverse Events [SAEs].

SECONDARY OUTCOMES:
Pharmacokinetics of JK06 | Day 1 of dosing through 7 days post last dose.
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics of JK06 | Day 1 of dosing through 7 days post last dose.
  Area Under the Curve (AUC)
Immunogenicity of JK06 by blood level measurement | Day 1 of dosing through 7 days post last dose.
  Lab draws at protocol defined intervals to measure Immunogenicity of circulating anti drug antibodies (ADA)
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression, assessed up to 104 weeks
  ORR according to RECIST v1.1.
Disease Control Rate (DCR) | "From date of randomization until the date of first documented progression, assessed up to 104 weeks
  The percentage of patients with a complete response, partial response, or stable disease for at least 2 consecutive tumor assessments.
Progression Free Survival (PFS) | "From date of randomization until the date of first documented progression, assessed up to 104 weeks
  Time from the date of initiation of study therapy to the date measurement criteria are first met for progressive disease or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Institut Jules Bordet, Brussels
  - UZ Ghent, Ghent
  - CHU UCL Namur - site Godinne, Yvoir
- Spain (4):
  - NEXT Oncology Barcelona, Barcelona
  - Vall d Hebron Institute of Oncology VHIO, Barcelona
  - Next Oncology Madrid, Madrid
  - START Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No